CLINICAL TRIAL: NCT02366507
Title: Systolic Blood Pressure Measurement in Critically-ill Patients
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Other Study IDs: BPD-02
Record Dates: First submitted 2014-07-25; First posted 2015-02-19 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2016-02

CONDITIONS: Hypotension; Shock
Keywords: hypotension; doppler; shock
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Traditional devices to measure blood pressure include automatic sphygmomanometer (pressure) cuff systems or manual blood pressures obtained by auscultation (listening with a stethoscope). Both these techniques fail to provide accurate and consistent blood pressure in the hypotensive (low blood pressure) state, which is often encountered in emergency departments and intensive care units. Alternately, invasive arterial pressure measurement is time-intensive, painful, expensive, and risks include bleeding, infection, and neurovascular injury.

In clinical practice, the Doppler velocimetry system is occasionally used in hypotensive, critically-ill patients when an immediate systolic blood pressure measurement is vital for clinical and therapeutic management. With a technique similar to that used to obtain a manual blood pressure, the Doppler velocimetry system can be used in place of the auscultation of the brachial pulse to accurately determine the systolic blood pressure. It is currently unknown whether additional information can be obtained by evaluation of the Doppler waveform in healthy vs. critically-ill patients. The goal is this project is to digitally record Doppler waveforms of critically-ill patients in the Emergency Department (ED) via a standard 8MHz (fetal) Doppler probe, correlate the Doppler readings with current blood pressure and heart rate, and determine if waveform shapes and parameters are predictive of hemodynamic compromise.

DETAILED DESCRIPTION:
Background/Significance:

Hypotension is common and predicts worse outcomes. Arterial hypotension, defined as an arterial systolic blood pressure (BP) less than 90 mmHg in adults, represents the hallmark of critical illness. Accurate arterial BP measurement is essential to deliver effective treatment, to guide resuscitation, and to assess interventions. Non-traumatic hypotension has been documented in as many as 19% of Emergency Department (ED) patients and those patients with hypotension have a 10-fold increased risk of sudden, unexpected in-hospital death.(1) Early hypotension is associated with increased mortality in survivors of cardiac arrest, stroke, and STEMI,(2-4) stressing the need for a tool to rapidly and accurately identify BP trends in order to effectively direct resuscitative measures. Additionally, Doppler waveforms may provide additional clues of impending hemodynamic deterioration before overt hypotension or shock ensues.

Disadvantages of the current system - The current initial standard for BP measurements in most hospitals is via an automated non-invasive BP device that uses oscillometric technology. This method has numerous limitations including non-continuous monitoring, missing or delays in identifying hypotensive episodes, inaccuracy or inability to measure BP due to various reasons including inaccurate cuff size or severity of hypotension. In one study, 34% of patients had a BP discrepancy of ≥ 20 mmHg with the oscillometric device compared to intra-arterial BP monitoring due to incorrect cuff size.(5) Oscillometric devices are sufficient for use in many clinical situations; however, notable exceptions include patients that are severely hypertensive, hypotensive, with arrhythmias, after trauma, and other critical clinical scenarios, whereby manual auscultatory BP measurement is preferred.(6) Even in non-critically ill patients, validation data of oscillometric measurements has been called into question.(7) The alternative to oscillometric devices is an intra-arterial catheter. Although accurate, intra-arterial catheters are invasive, technically difficult to insert, expensive, time-intensive, painful, and with risks including bleeding, infection, and neurovascular injury. Current guidelines for management of critically ill patients suggest intra-arterial BP measurement is preferred over automatic oscillometric non-invasive BP measurement. Despite this, in a recent survey of intensivists, 73% used non-invasive BP measuring devices in hypotensive patients.(8) For the above reasons, researchers have been investigating newer technology to replace the oscillometric technology; examples include Doppler and photoplethysmographic devices.(9;10) Newer technology- The research and application of Doppler technology for measuring BP is in its infancy and has yet to be fully realized. The benefits of such a device would include an accurate, non-invasive means to measure BP in critically-ill patients. Due the high-risk of missing hypotension, the possibility exists to commercialize the prototype for broader clinical use in non-critically ill patients as well. The accuracy of Doppler velocimetry is one important advantage. In an animal study comparing three indirect BP measuring instruments- a Doppler ultrasonic flowmeter, an oscillometric device, and a photoplethysmograph- to direct arterial pressure in cats, the Doppler and photoplethysmographic devices had the highest overall accuracy. (10) In clinical practice, when the initial automatic oscillometric BP device is unable to obtain a measurement due to hypotension, the manual Doppler technique is a common practice due to its reliability and referenced in one study as the "gold standard".(11) However, accurate systolic BP measurement is only one parameter of the device. The Doppler signal received from the arterial flow through the vessel has incredible potential to identify strength of pulse and other auditory queues. This has been well established in peripheral arterial disease, with descriptive terms used such as monophasic, biphasic, or triphasic pulses identified by Doppler. The novel device has the potential to identify a "sick" pulse as determined by changes in the Doppler waveform prior to hypotension ensues, as often, hypotension is very late in the course of the disease process. To date, there is no automatic sphygmomanometer/Doppler apparatus available.

This project will provide data to further the development of a novel blood pressure monitoring device that will enable non-invasive and near-continuous blood pressure monitoring and other hemodynamic information on critically-ill patients. Data from healthy volunteers using a standard 8MHz (fetal) Doppler probe have already been collected in a companion protocol in place at the University of North Carolina at Charlotte (UNCC).

Research Strategy:

1. Significance Identification of shock states before overt clinical evidence of shock (i.e., hypotension) is challenging. Determining whether Doppler-measured arterial waveforms can serve as a useful marker to identify hemodynamic compromise before shock ensues is unknown.
2. Approach Hypothesis: Doppler waveform patterns in critically-ill hypotensive patients have a unique and identifiable pattern.

Objectives:

1. Doppler waveforms will be collected from the brachial arteries of critically-ill patients that present to the ED with overt evidence of shock.

   This pilot study will allow us to obtain Doppler measurements in critically-ill patients for comparison to non-critically-ill patients collected previously in an IRB-approved study conducted at UNCC by the Co-PI.

   Doppler signal measurements will be obtained from 20 critically-ill patients with evidence of shock (i.e., hypotension with SBP < 90) in Emergency Department at Carolinas Medical Center. Eligible patients will be identified from the Code Sepsis clinical protocol alert by PCL currently utilized for other departmental studies or by direct report from the PI while working in the ED. Patients or a legally authorized representative will be approached for informed consent. The 8MHz Doppler probe, (fetal ultrasound probe), will be applied to the brachial artery, and the position adjusted until an adequate signal has been obtained. Doppler wave form data will be collected over the course of a few minutes. It is anticipated that the patients will experience minimal to no discomfort throughout this process.

   Expected technical difficulties and how we will overcome them: The technical difficulties will include ensuring consistent measurements, as the data will be collected by the investigators and clinical research staff.
2. Develop a computer algorithm that will distinguish "healthy" from "sick" Doppler waveforms.

Waveform characteristics from the ED patients will be compared to previously collected waveforms from normal volunteers. A computer algorithm will then be developed to identify distinguishing features between these waveforms (independent of blood pressure). We will use a similar power analysis as done by Holt et al.(11)

1. Algorithm Development: We will use MATLAB (The MathWorks, Inc) to analyze the Doppler signals obtained from the hypotensive/shock patients and compare them to prior obtained healthy patient data in order to identify unique wave characteristics of patients in shock.
2. Filtering: Optimum filtering software will be designed and perfected by the PIs, as required by the quantified audio piezo-electric signal, to determine most reliable and accurate Doppler waveform.

Sample Size Calculation Previous studies have used a power analysis that determined 18 observation sets (a set being one intra-arterial BP measurement and one Doppler BP measurement) to detect a difference of 10% (deemed clinically significant by investigators) between intra-arterial and Doppler BP with a SD for difference of 7.8 mmHg and an alpha of 0.05 using a two-sided one-sample t-test.

A power analysis was not performed for this pilot study. A sample size of twenty adult subjects (with Doppler recording during of < or = 5 minutes) was chosen to ensure sufficient observations. Further statistical techniques to improve association will be implemented as described in the initial prototype description.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Systolic Blood Pressure < 90 mmHg
3. Normotensive patients with SBP > or = 90 mmHg with suspected hypoperfusion/shock

Exclusion Criteria:

1. Patients < 18 years of age
2. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that present to the Emergency Department with hypotension or suspected shock.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
blood pressure measurements collected under standard of care | day 1
  blood pressure measurements collected under standard of care (manual or central line) will be used to compare to Doppler wave form readings.

CONTACTS AND LOCATIONS:
Overall Officials: David A Pearson, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States